CLINICAL TRIAL: NCT06371560
Title: Antibiotics, Antibiotic Resistance, and Prescribing Practices Among Periodontists: Cross Sectional Knowledge, Attitude and Practice (KAP) Study
Brief Title: Antibiotics, Antibiotic Resistance, and Prescribing Practices Among Periodontists: Cross Sectional KAP Study
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Attia, Lecturer, Cairo University
Other Study IDs: KAP-ABR-Perio
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Antibiotic Resistance; Antibiotic Use; Periodontitis
Keywords: KAP study; antibiotics use; antibiotic resistance; Prescribing practice; periodontal therapy; Periodontists
MeSH Terms: conditions — Periodontitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — online based questionnaire

SUMMARY:
Antibiotic resistance is a global health threats that require attention from all healthcare providers. In Periodontology, antibiotic is prescribed in many clinical situations. The aim of this study is to assess the followings among Periodontists (1) The knowledge, attitude, and practices (KAP) towards antibiotics and antibiotic resistance; (2) The prescribing practices of antibiotics in periodontal therapy; (3) The correlation between personal perception of antibiotics uses and the professional prescription patterns; and (4) The differences in antibiotics prescription in relation to the years of experience and the academic background.

DETAILED DESCRIPTION:
The study is designed as a cross-sectional online-based questionnaire, and it will be distributed among periodontitis. The study will be conducted in Egypt as a nationwide survey study. Google Form was used to develop online-based questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Periodontists who practice in Egypt.
* Must hold at least a master's degree in Periodontology
* Willing to provide informed consent to participate in the study and agree to use the data for publication purposes.

Exclusion Criteria:

* Periodontists who don not practice in Egypt.
* Periodontists who don not hold postgraduate degree

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population is representable sample of the periodontists who practice in Egypt and have postgraduate degree in Periodontology.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
KAP | 6 Months
  KAP on antibiotics and antibiotic resistance among periodontists

SECONDARY OUTCOMES:
The prescribing practices of antibiotics in periodontal therapy | 6 months
  how periodontists prescribe antibiotics in periodontal therapy
The correlation between personal perception of antibiotics uses and the professional prescription patterns | 6 months
  what is affect the antibiotic prescription by the periodontists
The differences in antibiotics prescription in relation to the years of experience and the academic background. | 6 months
  what is affect the antibiotic prescription by the periodontists

IPD SHARING:
Plan to Share IPD: Undecided
Any personal data will be protected and secured